CLINICAL TRIAL: NCT00333164
Title: Cilostazol-Aspirin Therapy Against Recurrent Stroke With Intracranial Artery Stenosis (CATHARSIS)
Brief Title: Cilostazol-Aspirin Therapy Against Recurrent Stroke With Intracranial Artery Stenosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Foundation for Biomedical Research and Innovation (Other); Neurology, Tokyo Women's Medical University, School of Medicine (Other); Kobe City General Hospital (Other); Tohoku University (Other); Kyushu University (Other); Department of Neurology, Saiseikai Central Hospital (Unknown); China National Center for Cardiovascular Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHA STROKE04-01
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2012-08

CONDITIONS: Cerebrovascular Disease
Keywords: intracranial arteriosclerosis; cilostazol; Platelete aggrigation inhibitors dual antiplatelet therapy; Drug therapy, combination; Clinical trials
MeSH Terms: conditions — Cerebrovascular Disorders; Intracranial Arteriosclerosis | interventions — Cilostazol

INTERVENTIONS:
Drug: Asprin, Cilostazol

SUMMARY:
Multi-center, open-labelled randomized controlled trial, to study the effect of aspirin plus cilostazol and aspirin alone on the progression of intracranial arterial stenosis, in 200 chronic stroke patients with 50-99% stenosis, to be followed up for 2 years

DETAILED DESCRIPTION:
Intracraial arterial stenosis (IAS) is more common in Asia, including Japanese, than in Cocasian. Also, stroke recurrence rate is high in patients with such lesions, despite medical treatment. Accoding to the result of WASID (N Engl J Med 2005;352:1305-16), warfarin is not recommended because of the concern of safety (higher risk of intracranial hemorrhage and death when compared with aspirin), wheras the efficacy of aspirin is not enough in symptomatic IAS patients. Under these conditions, we planned to conduct a nationwide multi-center, open labelled, randomized controlled trial to compare the effect of aspirin plus cilostazol (phosphodiestrase type 3 inhibitor) and aspirin alone on the progression of IAS in 200 IAS patients with ischemic stroke after 2 weeks to 6 months of onset. Patients are randomly allocated to either of two groups. Aspirin 100mg/day plus cilostazol 200 mg/day is given to the 100 patients in one group, and aspirin 100 mg/day alone is given to 100 patients in another group.

Follow-up period is at least two years. The primary endpoint is progression of IAS on MRA at two years after randomization. The secondary endpoints are cardiovascular events (ischemic stroke, myocardial infarct, and other vascular events), death, serious adverse events, new silent brain infarcts, and activity of daily life. The purpose of this study is to establish the best medical treatment in symptomatic IAS patients. This study will also provide important information for the future randomized controlled study to compare medical treatment alone and intravascular intervetnion (PTA and/or stenting) in these patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Ischemic stroke after two weeks to six months from onset,
* (2) Responsible lesion identified on MRI,
* ( 3) Intracranial arterial stenosis >50% on MRA in the territory of responsible lesion,
* (4) Intracranial arterial stenosis in suproclinoid internal carotid arterry, M1 portion of midlle cerebral artery, or basilar artery,
* (5) Age of 45 to 85 years,
* (6) Able to visit out-patient clinic, and
* (7) Written informed consent obtained from patient or family.

Exclusion Criteria:

* (1) Patients with potential cardiac embolic sources,
* (2) Patients receiving cilostazol,
* (3) Patients on warfarin treatment,
* (4) Patients in whom MRI cannot be perfomed,
* (5) Patients in whom PTA or bypass surgery is planned,
* (6) Patients with history of symptomatic intracranial hemorrhage, other hemorrhagic diseases (active peptic ulcer etc.), hemophilia or coagulation abnormalities,
* (7) Patients with hypersensitivity to cilostazol or aspirin,
* (8) Patients with congestive heart failure or uncontrollable angina pectoris,
* (9) Patients with thrombocytopenia (<100,000/mm3),
* (10) Patients with liver dysfunction (AST or ALT >100 IU/L),
* (11) Patients with renal dysfunction (Creatinin >2.0 mg/dl),
* (12) Patients who cannot to be followed up during the study period,
* (13) Patients who are enrolled in other clinical trials, and
* (14) Patients inadequate for this study by other reasons.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Progression of intracranial arterial stenosis after two years

SECONDARY OUTCOMES:
Cardiovascular events (ischemic stroke, cardiac infarctin, and other vascular events ）,
death (stroke death, vascular death except for stroke ）,
serious adverse events, new silent brain infarcts, and degrees of activity of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Uchiyama, M.D. PhD, Principal Investigator — Department of Neurology, Tokyo Women's Medical University School of Medicine; Nobuyuki Sakai, M.D. PhD, Principal Investigator — Kobe City General Hospital
Locations (1):
- Tokyo Women's Medical University School of Medicine, Shinjuku-ku, Tokyo, Japan